CLINICAL TRIAL: NCT00154557
Title: Influence of the Psychophysiological Status of Elite Judo Athletes on Their Performance and Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261701413
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2004-08

CONDITIONS: Injury
Keywords: Judo, Performance, Injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

INTERVENTIONS:
Behavioral: elite judo athletes program

SUMMARY:
Judo is one of the possible items in our country to win the first prize in Olympics. However, scientific research in this field is not enough to support the coaches to train the athletes. Series of research should be planned and executed to help the coaches and to promote the performance of our athletes. This is the first step of the serial research. The purposes of this study are: in the first year, to find the correlations between the physiological/psychological competitive abilities of the second/third year athletes and their performance/injury status. And, the physiological/ psychological competitive abilities of the first year athletes will be collected in the beginning of this year. And then, their performance/injury status will be followed through the whole year and to the end of the second year monthly. The purposes of this study in the second year are to find the causation of the physiological/ psychological competitive abilities in the first year with the performance/injury status in the second year.

The subjects of this study are from 4 senior high schools in the north part of Taiwan which performed well in national judo competition in senior high schools in the past years. The study designs are both cross-sectional and prospective. In the part of the second/third year athletes, it is a cross-sectional design, and in the part of the first year athletes, it is a prospective design. The physiological status will be assessed with their general fitness and balance. The fitness test includes body composition, strength, power, endurance, agility, coordination, balance, flexibility, and cardiopulmonary capacity. The psychological competitive abilities will be assessed with a questionnaire. Injury and the possible causes will also be collected with a questionnaire monthly. Finally, the data will be analyzed with descriptive analysis, chi-square test, t-test and regression analysis to show their characteristics, correlations and causations.

DETAILED DESCRIPTION:
Judo is one of the possible items in our country to win the first prize in Olympics. However, scientific research in this field is not enough to support the coaches to train the athletes. Series of research should be planned and executed to help the coaches and to promote the performance of our athletes. This is the first step of the serial research. The purposes of this study are: in the first year, to find the correlations between the physiological/psychological competitive abilities of the second/third year athletes and their performance/injury status. And, the physiological/ psychological competitive abilities of the first year athletes will be collected in the beginning of this year. And then, their performance/injury status will be followed through the whole year and to the end of the second year monthly. The purposes of this study in the second year are to find the causation of the physiological/ psychological competitive abilities in the first year with the performance/injury status in the second year.

The subjects of this study are from 4 senior high schools in the north part of Taiwan which performed well in national judo competition in senior high schools in the past years. The study designs are both cross-sectional and prospective. In the part of the second/third year athletes, it is a cross-sectional design, and in the part of the first year athletes, it is a prospective design. The physiological status will be assessed with their general fitness and balance. The fitness test includes body composition, strength, power, endurance, agility, coordination, balance, flexibility, and cardiopulmonary capacity. The psychological competitive abilities will be assessed with a questionnaire. Injury and the possible causes will also be collected with a questionnaire monthly. Finally, the data will be analyzed with descriptive analysis, chi-square test, t-test and regression analysis to show their characteristics, correlations and causations.

ELIGIBILITY:
Inclusion Criteria:

* senior high school student elite judo athletes

Exclusion Criteria:

-

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2004-08; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: J Y Tsauo, PhD, Study Director — Grad School of PT, College of Medicine, NTU
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan